CLINICAL TRIAL: NCT06425575
Title: Resolution of Pudendal Neuralgia in Chronic Pelvic Pain Using a Novel Biologic Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: The Cooper Health System (Other)
Responsible Party: Principal Investigator, Thomas N. Tulenko, Adjunct Professor, Thomas Jefferson University
Other Study IDs: 18D.719
Record Dates: First submitted 2024-02-21; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Chronic Pelvic Pain Syndrome
Keywords: pudendal neuralgia
MeSH Terms: conditions — Pudendal Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: Amniotic suspension allograft — the amniotic suspension allograft consists of fresh amniotic fluid into which micronized amniotic membrane has been added as a suspension.
  Other Names: Rheo, Flowgraft

SUMMARY:
This goal of this study is to determine whether a novel biologic, i.e., an "amniotic suspension allograft" (ASA) will reduce pain and improve quality of life (QoL) in women stricken with chronic pelvic pain (CPP). The main questions it aims to answer are:

* Weather pain in the genitalia is reduced with treatment
* Weather bladder or urination pain is reduced with treatment
* Weather any adverse events occur following treatment Patient responses to pain and QoL will be collected before and 6-12 months after treatment.

DETAILED DESCRIPTION:
This is an observational study and is driven by the hypothesis that novel biologic, i.e., an "amniotic suspension allograft" (ASA) will reduce pain and improve quality of life in women stricken with chronic pelvic pain (CPP). This clinical trial is performed in a hospital-based practice at Thomas Jefferson University in which all patients over the age of 18 presenting with clinically defined CPP will be accepted into the study and therefore all patients will be treated with the ASA; no patients with CPP will be excluded from the study. This small study is not funded so the patients will not be randomized and there will not be any "control" subjects receiving placebo instead of the ASA product. Upon arriving to the hospital, but just prior to treatment, all patients will be asked to fill out a consent form and a pre-procedure questionnaire regarding pain, discomfort and quality of life issues they've been experiencing prior to treatment. They will then be brought into the operating room, placed in the lithotomy position, and briefly anesthetized (15-30 min). Once anesthetized, the urogynecologist will feel for an opening in the pelvic bone (ischium) by inserting her fingers into the vagina. The opening (Alcock's canal) in the ischium exposes the pudendal nerve which carries pain signals from the vagina and nearby tissues to the brain's pain centers. Once the medial aspect of Alcock's canal is clearly identified by the doctor's fingers, a 6 inch pudendal trumpet needle will be advanced through the vaginal wall and guided and placed near the pudendal nerve in Alcock's canal. A solution of the ASA along with sterile saline and the anesthetic marcaine (5 cc total) will be injected so as to infiltrate the pudendal nerve with this mixture. Marcaine is used to help suppress any acute pain that may occur in the few hours after treatment. Both the left and right pudendal nerves will be thusly treated. When the patients awaken, they will receive a drink of choice and light snack like gram crackers or biscuits. When fully awake the patients will be allowed to leave the hospital accompanied with a companion, but not allowed to drive until the full effects of the anesthesia has worn off several hours later. From beginning to end, this procedure takes approximately one hour. To determine the extent to which any pain relief and quality of life have improved, or not, answers to a follow-up questionnaire will be solicited from each participating patient by telephone approximately 6 to 12 months after treatment. The questionnaire contains 14 questions addressing pain and discomfort, urination and impact of symptoms and takes about 10 minutes to compete. To protect patient privacy the data will be entered into an Excel spreadsheet with the patients' names replaced by a number and date of birth replaced with just their age. The data will be digitized, analyzed and statistical significance will be evaluated buy a biostatistician. This study has been approved by the institutional review board (protocol number: 18D.719) prior to beginning.

ELIGIBILITY:
Inclusion Criteria: All patients 18 years of age or older who present with chronic pelvic pain -

Exclusion Criteria:

1. Under 18 years of age
2. Malignancy defined as terminal -

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — All patients with clinically demonstrable chronic pelvic pain who are 18 years or older..
Study Population: All women presenting with chronic pelvic pain who are over 18 and without terminal disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Overall Pain and overall quality of life | Between 6 and 12 months after treatment
  Pain in structures of the genitalia, rectum and pain during sexual activity

SECONDARY OUTCOMES:
Bladder pain and urination frequency | Between 6 and 12 months after treatment
  Symptoms relating to interstitial cystitis
Adverse events | Between 6 and 12 months after treatment
  Zero pain relief

CONTACTS AND LOCATIONS:
Overall Officials: Thomas N Tulenko, PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferwson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No